CLINICAL TRIAL: NCT01211171
Title: COugh Among Hypertensive Patients Treated With Telmisartan, Who Had to Stop previoUs ACE-I Treatment Due to couGH
Brief Title: COugh Among Hypertensive Patients Treated With Telmisartan, Who Had to Stop previoUs ACE-I Treatment Due to couGH in Poland
Acronym: COUGH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14881; KL0910PL (Other: Company internal); 15379 - KL0910SK (Other: Company internal); GM.2009-04-06.0017 (Other: Company internal)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
Keywords: Cough; Telmisartan; Bradykinin; Tolerability
MeSH Terms: conditions — Hypertension; Cough | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Telmisartan (Kinzal/Pritor, BAY68-9291)

INTERVENTIONS:
Drug: Telmisartan (Kinzal/Pritor, BAY68-9291) — Patients treated with telmisartan tablets under the real-life setting. Dosing regimen customised to the needs of each participating patient according to the investigators assessment

SUMMARY:
In the light of ONTARGET and TRANSCEND studies results, it would be interesting to investigate the real-life telmisartan treatment tolerability. It is well known and accepted that the Real-life setting is much more adequate to reflect the antihypertensive and safety properties of the drug in comparison to the organized and scheduled setting of the clinical trial. Because there are not much data on the cough in relation to telmisartan, therefore it would we worth to observe the cough frequency and general treatment tolerance in patients treated with telmisartan, who had to stop their previous ACE-I treatment due to cough.

ELIGIBILITY:
Inclusion Criteria: - hypertension

* age > 18
* ACE-I related cough Exclusion Criteria: - Current treatment with telmisartan
* Cholestatic disorders and severe hepatic failure
* Allergy to telmisartan
* Pregnancy and lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic hypertensive patients with cough caused by the ACE-i regardless any other factors.
Sampling Method: Probability Sample
Enrollment: 2498 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cough frequency among telmisartan treated patients, who had to stop their previous ACE-I treatment due to cough | 4 months after initiation

SECONDARY OUTCOMES:
General tolerability and safety of telmisartan treatment among patients, who had to stop their previous ACE-I treatment due to cough | 4 months after initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland